CLINICAL TRIAL: NCT03461783
Title: Activated Carbon Interphase Effect on Biofilm and Total Bacterial Load: A Randomized Pilot Study
Brief Title: Activated Carbon Interphase Effect on Biofilm and Total Bacterial Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock Liden, DPM (Individual)
Responsible Party: Sponsor-Investigator, Brock Liden, DPM, Principal Invesigator, Liden, Brock, DPM
Organization: Liden, Brock, DPM (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Carbon Dressing
Record Dates: First submitted 2018-01-11; First posted 2018-03-12 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Zorflex Activated Carbon Dressing (Experimental): Patients randomized into the experimental group will only be treated using an activated carbon dressing (Zorflex® Activated Carbon Cloth Dressing; Chemviron Carbon Cloth Carbon, West Midlands, United Kingdom; a division of Calgon Carbon Corporation, Pittsburgh, PA) for wet wounds or with saline and Zorflex® Activated Carbon Cloth Dressing for dry wounds.
  Interventions: Device: Zorflex Activated Carbon Dressing
- Standard of Care for Wound Care (Active Comparator): Patients with wet wounds randomized into the control group will be treated using foam, calcium alginate or compressive dressings, whereas those with dry wounds will be treated with hydrogel and compressive dressings.
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Zorflex Activated Carbon Dressing — Antimicrobial dressing
  Arms: Zorflex Activated Carbon Dressing
Device: Standard of Care — foam, calcium alginate, hydrogel, or compressive dressings
  Arms: Standard of Care for Wound Care

SUMMARY:
The purpose of this randomized, prospective study is to evaluate how this activated carbon dressing affects the total bacterial load and biofilm in a wound bed in wounds of the lower extremity and foot. We anticipate that the use of Zorflex® Activated Carbon Cloth dressing will maintain the bacterial burden in the wound bed below the level of critical colonization, with potential secondary benefits of pain reduction, decrease in inflammation, and control of odor. Wound bed healing progression/acceleration also will be assessed.

DETAILED DESCRIPTION:
Wounds located on the lower extremity and feet are caused by several conditions, including diabetes and venous insufficiency. These types of wounds may not heal quickly and can become chronic. Chronic wounds are at risk for infection and limb amputation. As such, these wounds are a serious health issue, especially in diabetics and the elderly, and pose a significant public health burden. The healing of such wounds is an ongoing challenge to clinicians, who continue to seek effective management modalities.

The study treatment evaluated in this study is Zorflex® dressing (Chemviron Carbon Cloth Carbon, West Midlands, United Kingdom; a division of Calgon Carbon Corporation, Pittsburgh, PA). According to the Instructions for Use for the product, it is a low-adherent, 100% pure activated carbon cloth dressing that highly conforms to the body contours and maintains contact with the wound surface. It provides an effective antimicrobial barrier for a minimum of 7 days per dressing, protecting the wound from invasive microorganisms, while exhibiting an antimicrobial effect against microorganisms already present in the wound. The dressing may be used either dry or moistened with sterilized water. Zorflex® is indicated as an antimicrobial dressing over dry or discharing, partial and full thickness wounds.

The following unique properties of the activated carbon dressing are believed to aid in wound healing and patient comfort when used for wound management: 1) antimicrobial; 2) odor management; and 3) conductive. The dressing is antimicrobial and manages odor because of its naturally occurring "van der Waal's" electrostatic forces. These forces draw small gas or liquid molecules, including endotoxins and odor molecules, away from the wound into the highly structured micropores of the dressing, where they become trapped. Bacteria cells also are attracted to the dressing, but are too big to enter the micropores. Instead, the microorganisms become trapped on the surface, away from the wound bed. Electrostatic tension builds up in the trapped microorganisms until the tension overcomes the tensile strength of the cell walls, at which time the cell walls of the microorganisms rupture, killing the microorganisms. Any endotoxins released in the process are drawn into the micropores and also become trapped. The conductive nature of the dressing restores the body's natural transepithelial potential across the wound bed, thereby aiding in healing. The positive effects of electrostimulation on wound healing have been previously established.

Several studies, primarily case series, have reported promising preliminary results with the use of Zorflex® as an antimicrobial dressing for wound management. In a case series involving four patients with recalcitrant venous leg ulcers that were prone to recurrent infection, treatment with this particular activated carbon cloth dressing resulted in a reduction in clinical signs of infection, such as exudate and pain levels, and improvement in wound bed appearance after 7 days. A retrospective study evaluating the use of this activated carbon cloth dressing for the management of 18 chronic wounds demonstrated 90.7% wound closure at 5 weeks. Finally, another case series examining the use of Zorflex® in chronic lower extremity and foot wounds demonstrated a reduction in odor control and progression of healing with the use of the dressing.

Studies examining the efficacy of such activated carbon dressings are limited and, therefore, more research, particularly randomized and prospective in design, is needed to better elucidate possible effects of this dressing on preventing infection and promoting healing. The purpose of this multi-center, randomized, prospective study is to evaluate how this activated carbon dressing affects the total bacterial load and biofilm in a wound bed in wounds of the lower extremity and foot. We anticipate that the use of Zorflex® Activated Carbon Cloth dressing will maintain the bacterial burden in the wound bed below the level of critical colonization, with potential secondary benefits of pain reduction, decrease in inflammation, and control of odor. Wound bed healing progression/acceleration also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age.
* Patients of both genders and all races.
* Patients who are in good general health.
* Patients with ankle-brachial index (ABI) measurements greater than 0.5.
* Patients with full-thickness lower extremity diabetic or venous wounds that are not currently being treated with antimicrobial products.
* Patients with full-thickness wounds that are not yet extending to the bone or tendon.
* Patients with wounds present for at least 4 weeks, but no longer than one year.
* Patients with initial bacterial load greater than or equal to 104 colony forming units (CFUs), but less than or equal to 106 CFUs.
* Patients who have voluntarily signed the informed consent form, including HIPAA Authorization.

Exclusion Criteria:

* Patients who are younger than 18 years of age.
* Patients with autoimmune conditions.
* Patients with ABI measurements less than 0.5 or with lower extremities that are non-interventional or by-passable.
* Patients with full-thickness lower extremity pressure wounds.
* Patients with diabetic or venous wounds that are being treated with antimicrobial products.
* Patients with full-thickness wounds with exposed bone or tendon.
* Patients with wounds present less than 4 weeks or one year or longer.
* Patients with ulcers that had an initial bacterial load less than 104 CFUs or greater than 106 CFUs.
* Patients who are pregnant or lactating.
* Patients with known allergy(ies) to any of the components of the study dressing.
* Patients who are considered by the investigator for any reason to be an unsuitable candidate.
* Patients who are unwilling or unable to follow the follow-up evaluation schedules.
* Patients who refuse to voluntarily sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Total Bacterial Load | 4 weeks
  Total bacterial load will be measured total colony forming units (CFUs) as determined from laboratory findings

SECONDARY OUTCOMES:
Pain Associated with Wound | 4 weeks
  Patients will rate their pain on a Visual Analog Scale (VAS) that consists of a 10cm (100mm) line with the descriptor "no pain" positioned at the left pole and the descriptor "worst pain imaginable" positioned at the right pole.
Wound Bed Inflammation | 4 weeks
  Protease laboratory measurements of the wound bed will be use to elevate wound bed inflammation.
Wound Odor | 4 weeks
  Wound odor will be assessed by both the patient and investigator using Visual Analog Scale (VAS) that consists of a 10cm (100mm) line with the descriptor "no odor" positioned at the left pole and the descriptor "extremely offensive odor" positioned at the right pole.
Wound Size Progression | 4 weeks
  Wound size measurements obtained from the software utilized by the eKare inSight™ (eKare, Inc., Fairfax, VA) system will be used to determine wound bed healing progression.

CONTACTS AND LOCATIONS:
Overall Officials: Brock Liden, DPM, Principal Investigator — Circleville Foot & Ankle LLC
Locations (2):
- United States (2):
  - Circleville Foot & Ankle, LLC, Circleville, Ohio
  - Hocking Valley Community Hospital, Logan, Ohio

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Isseroff RR, Dahle SE. Electrical Stimulation Therapy and Wound Healing: Where Are We Now? Adv Wound Care (New Rochelle). 2012 Dec;1(6):238-243. doi: 10.1089/wound.2011.0351. PMID 24527312
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Kalinski CK, Schnepf M, Laboy D, Hernandez L, Nusbaum J, McGrinder B, Comfort C, Alvarez OM. Effectiveness of a Topical Formulation Containing Metronidazole for Wound Odor and Exudate Control. Wounds. 2005;17(4):84-90.
- [Background] Miller MS, Markey L, Yoder R. A link to reducing the stink - use of a unique carbon based textile dressing Zorflex® to promote healing while significantly reducing wound odor in diabetic and venous ulcers - a case series of three. Presented as a poster at the Wild on Wounds (WOW) National Wound Conference, Las Vegas, NV, Aug 31-Sept 3, 2016.
- [Background] Murphy N. Reducing infection in chronic leg ulcers with an activated carbon cloth dressing. Br J Nurs. 2016 Jun 23;25(12):S38-44. doi: 10.12968/bjon.2016.25.12.S38. PMID 27345081
- [Background] Young S, Gray S, and Hampton S. A retrospective study to evaluate the effect of an activated carbon dressing on chronic wounds. Presented as an e-poster at the 2016 European Wound Management Association (EWMA), Bremen, Germany, May 11-13, 2016.
- [Background] Zorflex® Instructions for Use. http://zorflex.com/what-is-zorflex/, accessed on January 17, 2017.